CLINICAL TRIAL: NCT00875576
Title: Influence of Parents and Friends on Children and Adolescents
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Responsible Party: Sarah-Jeanne Salvy, Ph.D., University at Buffalo
Other Study IDs: DB# 2354
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2009-04

CONDITIONS: Healthy
Keywords: social influences; meals; obesity; amount of food consumed
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to directly compare the effects of parents and friends on overweight and non-overweight children and adolescents' food intake and food selection using a cross-sectional design. Overweight and non-overweight children (5-6 year-old) and adolescents (13-14 year-old) will share a meal with a friend and with a parent on separate occasions. Participants' food selection and the amount of food they consumed will be compared across conditions.

Hypothesis 1: The investigators hypothesize that overweight children and adolescents will select more unhealthy food items and eat more in the presence of an overweight friend than when eating with a lean friend; whereas lean participants eating with an overweight friend will eat a similar amount of food than lean youth eating with a lean friend.

Hypothesis 2: The investigators predict that overweight children and adolescents (but not lean children and teens) will consume more food in the presence of their mother than in the presence of a friend.

Hypothesis 3: The investigators also predict that overweight youth's energy intake will be related to parental prompts.

Hypothesis 4: The investigators expect greater similarities in terms of food selection and food intake between adolescents and their friend than between adolescents and their parent.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls ages 5-6 yrs and 12-14 yrs and their mothers
* Children must have a BMI greater than or equal to 15th percentile for their age
* Children and their mothers must have at least a moderate liking of the study foods used

Exclusion Criteria:

* Participants should not have any food allergies
* Participants should have no dietary restraints
* Participants should have no psychopathology that can limit food choice and alter eating
* Participants should have no developmental disabilities that can limit food choice and alter eating
* Participants cannot have a cold or upper respiratory distress that could influence taste, appetite or olfactory sensory responsiveness
* Participants cannot be on any medications that could influence taste, appetite or olfactory sensory responsiveness

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Boys and girls ages 5-6 yrs and 12-14 yrs and their mothers.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
amount of food consumed | Measured once with a friend and once with a mother, both occurring within a week of each other.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Salvy, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Division of Behavioral Medicine, Buffalo, New York, United States

REFERENCES:
- [Derived] Salvy SJ, Elmo A, Nitecki LA, Kluczynski MA, Roemmich JN. Influence of parents and friends on children's and adolescents' food intake and food selection. Am J Clin Nutr. 2011 Jan;93(1):87-92. doi: 10.3945/ajcn.110.002097. Epub 2010 Nov 3. PMID 21048059